CLINICAL TRIAL: NCT04596995
Title: An Open-Label Extension Study to Investigate the Long-Term Safety, Tolerability, and Efficacy of Rozanolixizumab in Study Participants With Persistent or Chronic Primary Immune Thrombocytopenia (ITP)
Brief Title: A Study to Investigate the Long-term Safety, Tolerability, and Efficacy of Rozanolixizumab in Study Participants With Persistent or Chronic Primary Immune Thrombocytopenia (ITP)
Acronym: myOpportunITy3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic Business Decision; Not a safety decision
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP0004; 2019-000883-40 (EudraCT Number)
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: ITP; UCB7665; Rozanolixizumab; Primary immune thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — rozanolixizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rozanolixizumab Treatment Arm (Experimental): All study participants will receive fixed-unit doses of rozanolixizumab across body weight tiers at pre-specified time points during the Treatment Period. Doses will be adjusted based on platelet count values or medical needs.
  Interventions: Drug: Rozanolixizumab

INTERVENTIONS:
Drug: Rozanolixizumab — Study participants receive rozanolixizumab by subcutaneous infusion during the Treatment Period.
  Other Names: UCB7665

SUMMARY:
The purpose of this study is to assess the long-term safety, tolerability and clinical efficacy of treatment with rozanolixizumab.

ELIGIBILITY:
Inclusion Criteria:

* Study participant completed TP0003 [NCT04200456] or TP0006 [NCT04224688] until Visit 27 (Week 25) and, in the opinion of the investigator, has been compliant with the TP0003 or TP0006 study assessments
* The study participant is considered reliable and capable of adhering to the protocol, visit schedule, or medication intake according to the judgment of the investigator
* Study participants may be male or female:

  1. A male participant must agree to use contraception during the Treatment Period and for at least 3 months after the final dose of study treatment and refrain from donating sperm during this period
  2. A female participant is eligible to participate if she is not pregnant as confirmed by a negative urine pregnancy test and not planning to get pregnant during the participation in the study, not breastfeeding, and at least one of the following conditions applies:

Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow the contraceptive guidance during the Treatment Period and for at least 3 months after the final dose of study treatment

Exclusion Criteria:

* Study participant has any ongoing investigational medicinal product (IMP)-related serious adverse event (SAE) or ongoing severe IMP-related treatment-emergent adverse event (TEAE) experienced during TP0003 or TP0006
* Study participant has, at last available assessment of TP0003 or TP0006, 3.0x upper limit of normal (ULN) of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (27):
- Tp0004 50243, Boston, Massachusetts, United States
- China (3):
  - Tp0004 20179, Fuzhou
  - Tp0004 20185, Jinan
  - Tp0004 20194, Wuxi
- Tp0004 20050, Tbilisi, Georgia
- Tp0004 40369, Berlin, Germany
- Hungary (2):
  - Tp0004 40202, Győr
  - Tp0004 40178, Nyíregyháza
- Tp0004 40208, Florence, Italy
- Tp0004 20039, Iruma-gun, Japan
- Tp0004 20051, Chisinau, Moldova
- Poland (4):
  - Tp0004 40218, Gdansk
  - Tp0004 40222, Skorzewo
  - Tp0004 40219, Słupsk
  - Tp0004 40223, Warsaw
- Russia (2):
  - Tp0004 20052, Moscow
  - Tp0004 20053, Saint Petersburg
- Tp0004 40268, Madrid, Spain
- Taiwan (2):
  - Tp0004 20095, Taipei
  - Tp0004 20099, Taipei
- Ukraine (6):
  - Tp0004 20061, Cherkasy
  - Tp0004 20060, Dnipropetrovsk
  - Tp0004 20062, Ivano-Frankivsk
  - Tp0004 20063, Kyiv
  - Tp0004 20064, Kyiv
  - Tp0004 20100, Zaporizhzhia
- Tp0004 40234, Plymouth, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in January 2021 and completed prematurely in December 2022. Study participants from TP0003 (NCT04200456) or TP0006 (NCT04224688) who had completed the 24-week Treatment Period (irrespective of rescue therapy) and met eligibility criteria for TP0004 were enrolled in this study.
Pre-assignment Details: Participant Flow refers to the Enrolled Set.
Groups:
- Rozanolixizumab: In TP0004, participants received a fixed unit dose of rozanolixizumab subcutaneous (sc) infusion at the assigned dose level in the parent studies (TP0003 and TP0006), for one year, starting from Day 1 (which corresponds to Week 25 of the parent studies). The dose of rozanolixizumab could be increased or decreased based upon the platelet count and across body weight tiers.
Period: Overall Study
Arm/Group | Rozanolixizumab
Started | 43
Completed | 14
Not Completed | 29
Not completed — Lack of Efficacy | 8
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 12
Not completed — Sponsor decision | 3
Not completed — Enrolled in managed access program | 3

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to Enrolled Set which consisted of all study participants who signed the informed consent form (ICF).
Groups:
- Rozanolixizumab: In TP0004, participants received a fixed unit dose of rozanolixizumab sc infusion at the assigned dose level in the parent studies (TP0003 and TP0006), for one year, starting from Day 1 (which corresponds to Week 25 of the parent studies). The dose of rozanolixizumab could be increased or decreased based upon the platelet count and across body weight tiers.
Arm/Group | Rozanolixizumab
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (13.7)
Age, Customized [Count of Participants; unit: Participants]
  18 - <65 years | 41
  >=65 - <85 years | 2
  >=85 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8
  White | 33
  Other or Mixed | 1
  Missing | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to the IMP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP. TEAEs are defined as AEs starting after the time of first IMP administration up to and including 8 weeks (56 days) after the final dose.
Time Frame: From Baseline to end of Safety Follow-Up Period (up to Week 60)
Population: Safety Set included all study participants who received at least 1 dose of IMP (partial or full).
Measure: Number; unit: percentage of Participants
Arm/Group | Rozanolixizumab
Number analyzed (Participants) | 43
percentage of Participants | 90.7

2. Primary Outcome: Percentage of Participants With TEAEs Leading to Permanent Withdrawal of Rozanolixizumab (ie, Study Discontinuation)
Description: as for outcome 1
Time Frame: From Baseline to end of Safety Follow-Up Period (up to Week 60)
Population: Safety Set included all study participants who received at least 1 dose of IMP (partial or full).
Measure: Number; unit: percentage of Participants
Arm/Group | Rozanolixizumab
Number analyzed (Participants) | 43
percentage of Participants | 0

3. Secondary Outcome: Percentage of Participants With Stable Clinically Meaningful Response Without Rescue Therapy at ≥70% of the Visits Over the Planned 52-week Treatment Period Starting at Week 4
Description: Stable Clinically Meaningful Response was defined as Clinically Meaningful Response (ie, platelet count ≥50×10^9/L) without rescue therapy at ≥70% of the visits over the planned 52-week Treatment Period starting at Week 4.
Time Frame: Over the 52-week Treatment Period (starting at Week 4)
Population: Safety Set included all study participants who received at least 1 dose of IMP (partial or full).
Measure: Number; unit: percentage of participants
Arm/Group | Rozanolixizumab
Number analyzed (Participants) | 43
percentage of participants | 16.3

4. Secondary Outcome: Change From Baseline in Immune Thrombocytopenia-Patient Assessment Questionnaire (ITP-PAQ) to Week 53 or 55 Symptoms Domain Score
Description: The ITP-PAQ Version 1 is a 44 item disease-specific Health-Related Quality of Life questionnaire developed for use in adults with chronic ITP. It includes 10 scales, Four of the scales measure physical health: Symptoms (6 items), Bother (3 items), Fatigue (4 items), and Activity (2 items). Two of the scales measure emotional health: Fear (5 items) and Psychological (5 items) Health. The remaining four scales measure other aspects of quality of life (QOL): Work QOL (4 items), Social QOL (4 items), Women's Reproductive QOL (6 items) and Overall QOL (5 items). Each item is rated on a Likert-type scale containing 4 to 7 responses. All item scores are transformed to a 0 to 100 continuum and are weighted equally to derive individual scale scores and the total score (0-100) is calculated as per the formula: Sum of item scores within the scale/raw sum range*100. Higher scores indicate better health status.
Time Frame: Week 53 or 55, compared to Baseline
Population: Safety Set included all study participants who received at least 1 dose of IMP (partial or full). Here, number of participants analyzed signifies those who were evaluable for this outcome measure and number analyzed signifies participants who were evaluable at specified time points. Week 53 was used for study participants who finished the study on weekly dosing, and Week 55 was used for study participants who finished the study on biweekly dosing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rozanolixizumab
Number analyzed (Participants) | 12
score on a scale
  Week 53: number analyzed (Participants) | 7
  Week 53 | 2.98 (11.21)
  Week 55: number analyzed (Participants) | 5
  Week 55 | 4.17 (12.50)

ADVERSE EVENTS:
Time Frame: From Baseline to end of Safety Follow-Up Period (up to Week 60)
Description: Treatment-emergent AEs are defined as AEs starting after the time of first investigational medicinal product (IMP) administration up to and including 8 weeks (56 days) after the final dose. TEAEs were analyzed for Safety Set.
Arm/Group | Rozanolixizumab
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 9/43
Other Adverse Events (participants affected / at risk) | 31/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rozanolixizumab (N=43)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (2)
Haemorrhage (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rozanolixizumab (N=43)
Anaemia (Blood and lymphatic system disorders) | 3 (11)
Diarrhoea (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 5 (9)
Vomiting (Gastrointestinal disorders) | 3 (7)
Fatigue (General disorders) | 5 (6)
Pyrexia (General disorders) | 9 (26)
COVID-19 (Infections and infestations) | 7 (8)
Pharyngitis (Infections and infestations) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Body temperature increased (Investigations) | 5 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 18 (58)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT04596995/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT04596995/SAP_001.pdf